CLINICAL TRIAL: NCT04504617
Title: A Theory-based Nutrition Education Intervention to Enhance Complementary Feeding Practices Among Young Children in Southern Ethiopia
Brief Title: Nutrition Education Intervention to Enhance Complementary Feeding Practices Among Infants in Southern Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas Tech University (Other)
Collaborators: Kansas State University (Other); Hawassa University (Other)
Responsible Party: Principal Investigator, Mary Murimi, Professor of Nutrition, Texas Tech University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB2019-664
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Infant Malnutrition
Keywords: Infant undernutrition; Complementary feeding
MeSH Terms: conditions — Infant Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will consist of six kebeles with a total of 90 pairs of mothers and their children that will receive the nutrition education intervention to enhance complementary feeding practices first. The six lessons will be delivered in a period of 6 weeks. Before the intervention this groups will be assessed with the baseline assessment. After the intervention, this group will be assessed in three time points (post-intervention, follow-up 1 and follow-up 2).
  Interventions: Behavioral: Nutrition education intervention to enhance complementary feeding practices
- Delayed Intervention Group (Active Comparator): This arm will consist of the six kebeles with a total of 90 pairs of mothers and their children that will not receive the intervention immediately. This group will first complete the baseline and the second assessment. After the second assessment, this group will receive the nutrition education intervention to enhance complementary feeding practices. After the intervention, this group will be assessed in two additional time points (post-intervention and follow-up 1).
  Interventions: Behavioral: Nutrition education intervention to enhance complementary feeding practices

INTERVENTIONS:
Behavioral: Nutrition education intervention to enhance complementary feeding practices — The intervention consist of a six-week nutrition education intervention developed following the DESIGN procedure and the Socio-Cognitive Theory. The intervention consisted of six three-hour weekly sessions that covered topics such as 1) importance and benefits of exclusive and continuing breastfeeding; 2) nutrition for lactating mothers; 3) importance and benefits of complementary feeding practices; 4) risks for starting complementary feeding too early or too late; 5) complementary feeding practices for each age group (6-8, 9-11, and 12-24); 6) importance and benefits of dietary diversity; 7) importance of animal-source foods; 8) importance and benefits of following water, sanitation, and hygiene practices; 9) food safety practices when preparing meals; and 10) the recommended hand-washing protocol. Each lesson was designed to provide a lecture, a discussion using counseling cards, a cooking demonstration with tasting session, and key messages.

SUMMARY:
Child undernutrition is a worldwide public health problem that has persisted in African countries. For instance, the most recently reported prevalence rates of stunting (38%), underweight (24%), and wasting (10%) among children under the age of five in Ethiopia is higher than the global prevalence. The causes of undernutrition are classified in the following manner: immediate causes, such as inadequate dietary intakes; underlying causes, such as household food insecurity and inadequate care and feeding practices; and basic causes, which involve the household's inadequate access to education, employment, and income, among others. Evidence has demonstrated that nutrition education interventions (NEI) may influence both underlying and immediate causes of child undernutrition. For instance, nutrition education interventions have the potential of preventing the underlying causes of child undernutrition by improving mothers' knowledge in care and feeding practices, and further improving the quality and quantity of dietary intake, which is considered an immediate cause of child undernutrition. Moreover, nutrition education interventions designed to improve infant and young child feeding (IYCF) practices, such as dietary diversity, frequency, and adequacy, are considered a high impact strategy that may substantially reduce stunting. Preliminary data from Hawassa University (collaborating institution in this project) demonstrated that approximately 86% of the children residing in Arsi Negele, Wondo Genet, and Dale districts in Oromia and Southern Nations, Nationalities and Peoples' (SNNP) regions in Ethiopia do not receive adequate complementary feeding practices. Such lack of optimal complementary feeding practices may compromise a child's growth, development, and survival. Therefore, there is a critical need for improving child complementary feeding practices to promote their well-being and adequate nutritional status. Thus, the main purpose of this study is to improve child feeding practices and related nutritional status by improving the mother's knowledge, attitudes, and practices (KAP) of complementary feeding practices for their children aged six to 23 months in three woredas located in Oromia and SNNP. It is hypothesized that after the NEI mothers will improve their children' dietary diversity, frequency and adequacy.

DETAILED DESCRIPTION:
Elegibility criteria: residents that have lived in Arsi Negele, Wondo Genet, and Dale districts for at least one year, households that have children between 6 and 23 months of age, households where the mother is permanently presents, and households that speak sidamo or oromio.

Exclusion criteria: residents that have lived in Arsi Negele, Wondo Genet, and Dale districts for less than one year, households that have children under 6 months or above 23 months of age, households where the mother is not present, and households that do not speak sidamo.

Outcomes of this study are child feeding practices knowledge, attitudes, dietary diversity score, meal frequency score, adequacy diet score, continuing breastfeeding, maternal dietary diversity, and prevalence of stunting, wasting, and underweight.

ELIGIBILITY:
Inclusion Criteria:

* Infant that live in a household that has reside in Arsi Negele, Wondo Genet, and Dale districts for at least one year
* Infants that are within the age of 6 to 23 months at the time of the recruitment
* Infants that live in households where the mother is permanently present
* Infants that live in a household where the mother speaks sidamo or oromio.

Exclusion Criteria:

* Infants that live in a household that has reside in Arsi Negele, Wondo Genet, and Dale districts for less than one year
* Infants that are under 6 months or above 23 months of age at the time of the recruitment
* Infants that live in households where the mother is not present
* Infants that live in households where the mother does not speak sidamo or oromio
* Infants that have an illness that require a special nutrition treatment

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Dietary diversity score | Six weeks
  The dietary diversity score will be measured using the population indicator of minimum dietary diversity score for children aged 6 to 23 months designed by The Who. This measurement assess the consumption of seven food groups through seven yes-no questions. The food groups that are assessed are the following: 1) grains, roots and tubers; 2) legumes and nuts; 3) dairy products (milk, yogurt, cheese); 4) flesh foods (meat, fish, poultry, and organ meats); 5) eggs; 6) vitamin A rich fruit and vegetables; and 7) other fruits and vegetables. The total dietary diversity score for each participant will be the sum of the food groups that were responded with a yes answer. The maximum score possible is seven.
Meal frequency | Six weeks
  The meal frequency of children will be measured using a question that forms part of the Infant Young and Child Feeding Practices questionnaire provided by the WHO. This question assess the number of times that a baby had meals or snacks, other than liquids, through a multiple answer questions. The participating mother has the option to select the meal frequency from one to six times. The average meal frequency will be calculated for those breastfed and non-breastfed children.
Acceptable diet score | Six weeks
  This is an indicator that measures the proportion of children aged 6 to 23 months of age who receive the minimum feeding frequency and minimum dietary diversity. The acceptable diet score will be calculated using the proportion of children that meet the minimum dietary diversity and the minimum meal frequency divided by the total number of children. This score will be calculated for breastfed and non-breastfed children.

SECONDARY OUTCOMES:
Child feeding knowledge score | six weeks
  The child feeding knowledge score will be assessed using the questions obtained from the FAO Guidelines for assessing nutritional-related knowledge, attitudes, and practices. The section of knowledge includes 7 open-ended questions in which the data collector will ask an open-ended question to the mother and the mother will have to provide a short answer in her own words. The knowledge score per participant will be calculated based on the number of correct answers provided and an average score of participants will be calculated.
Child feeding maternal attitude score | six weeks
  The child feeding maternal attitude score will be assessed using the questions obtained from the FAO Guidelines for assessing nutritional-related knowledge, attitudes, and practices. The section of attitudes includes 7 three-point Likert scale questions. These questions will assess self-confidence, perceived benefits and barriers for providing diversity foods, frequently meals, and continued breastfeeding for their children aged 6 to 23 months. Responses will be codified to calculate an attitude score per participant. Responses will be codified in the following way: "no confident", "not good" and "challenging" as one; "ok/so-so", "you're not sure", and so-so as two; and "good" and "not challenging" as three.
Maternal dietary diversity score | six weeks
  The dietary diversity score will be measured using the Minimum Dietary Diversity for Women (MDD-W). This measurement assess the consumption of 10 food groups through 17 yes-no questions. The food groups that are assessed are the following: 1) grains, white roots, tubers, and plantains; 2) pulses (beans, peas, and lentils); 3) nuts and seeds; 4) dairy; 5) meat, poultry and fish; 6) eggs; 7) dark green leafy vegetables; 8) other vitamin-A rich fruits and vegetables; 9) other vegetables; and 10) other foods. The total dietary diversity score for each participant will be the sum of the food groups that were responded with a yes answer. The maximum score possible is ten.
Nutritional status | six weeks
  WHO Anthro software will be utilized to calculate weight-for-height z-score (WHZ), height-for-age z-score (HAZ), and weight-for-age z-score (WAZ). Then those children that have a -2 standard deviation in their WHZ, HAZ, and WAZ will be categorized as having wasting, stunting, or underweight. The prevalence of these nutritional status categories will be compared before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mary W Murimi, PhD, Principal Investigator — Texas Tech University
Locations (1):
- Hawassa University, Awasa, Southern Nations, Nationalities, and Peoples' Region, Ethiopia

IPD SHARING:
Plan to Share IPD: No